CLINICAL TRIAL: NCT06177392
Title: VARC-TAVI (VASCULAR CONTROL in TRANSCATHETER AORTIC VALVE IMPLANTATION)
Brief Title: VARC-TAVI VALVE IMPLANTATION)
Acronym: VARC-TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Daniel Tébar Márquez, Doctor of medicine, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VARC-TAVI 6571-2023.735
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Severe Aortic Stenosis; TAVI(Transcatheter Aortic Valve Implantation); Vascular Complications
Keywords: RADIAL ACCESS; RADIAL SECONDARY ACCESS; TAVI; SEVERE AORTIC STENOSIS; VASCULAR COMPLICATIONS; VARC-3
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RADIAL (Experimental): RADIAL ARTERY ACCESS AS SECONDARY ACCESS IN TAVI PROCEDURE
  Interventions: Procedure: Secondary TAVI access
- FEMORAL (Active Comparator): FEMORAL ARTERY ACCESS AS SECONDARY ACCESS IN TAVI PROCEDURE
  Interventions: Procedure: Secondary TAVI access

INTERVENTIONS:
Procedure: Secondary TAVI access — The randomization will determine whether radial or femoral artery puncture will be employed as the secondary access in the TAVI procedure.

SUMMARY:
SUMMARY:

The investigators are planning a clinical study to compare two methods of performing a procedure called TAVI, used in patients with severe aortic stenosis. In this procedure, the aortic valve is replaced in a less invasive way. Traditionally, access through the groin (femoral) is used, but now radial access (through the wrist) is being considered as an alternative.

Reasons for the Study:

* Currently, there is not enough solid evidence to support the choice between these two accesses.
* The investigators want to understand if radial access could be safer and have fewer complications compared to femoral access.

What the Investigators Will Measure:

* Major complications, such as bleeding or vascular injuries.
* Other important outcomes, such as functional recovery and quality of life.

How the Investigators Will Do It:

* The investigators will randomize patients to receive radial or femoral access.
* The investigators will record which type of access is used and assess complications and outcomes.
* The investigators will compare the results to understand if there are significant differences between the two groups.

Ultimate Goal:

* The investigators aim to improve the safety and efficacy of this procedure for patients.
* The results of this study will help doctors make informed decisions on how to perform TAVI.

Conclusion:

- This study is crucial for enhancing care for patients with aortic stenosis and ensuring the procedure is performed in the safest and most effective manner. The results will benefit patients and guide doctors in choosing the best approach for each individual.

DETAILED DESCRIPTION:
INTRODUCTION:

The TAVI procedure has been established as a safe and effective alternative for aortic valve replacement in patients with severe aortic stenosis. Vascular access plays a crucial role during the TAVI procedure, allowing the introduction of necessary devices for valve implantation, as well as protection and resolution of potential complications. Traditionally, femoral access has been the preferred approach for both main access (through which the valve navigates) and secondary access (serving as a guide during implantation and protection of the main access) due to its familiarity and technical ease. However, in recent years, radial access has gained popularity due to its theoretical potential to reduce vascular complications and improve participant recovery and quality of life. In this study, the investigators aim to demonstrate if there are differences between radial and femoral secondary access in transfemoral TAVI implantation.

JUSTIFICATION:

Conducting a clinical trial comparing radial and femoral secondary access in transfemoral TAVI implantation is crucial for several fundamental reasons. The main aspects supporting the need for such a clinical trial are outlined below.

1. Limited and Heterogeneous Evidence:

   * Observational studies and retrospective data supporting radial access as contralateral access during TAVI implantation exist, but they are non-randomized and subject to biases and methodological limitations. Prospective and controlled clinical trials are required to generate solid and reliable evidence.
2. Differences in Complication Rates:

   * Multiple clinical trials have shown a reduction in both vascular and non-vascular complications, major and minor, with radial access compared to femoral access in coronary catheterizations, even demonstrating a reduction in mortality. Similarly, observational studies suggest a similar trend for femoral and radial access as secondary access in TAVI, but these studies have multiple biases. A clinical trial would provide higher-level evidence regarding the existence of differences in vascular complications associated with the procedure.
   * Bleeding and Transfusions: Bleeding is a common complication after TAVI and is associated with increased morbidity and mortality. Several studies have demonstrated a reduction in bleeding and the need for transfusions in TAVI participants with radial access compared to femoral access.
   * Other Complications: Meta-analyses of observational studies have also observed a reduction in peri-procedural renal failure and stroke in participants with radial access. However, due to study limitations, other variables may influence these observations, requiring evaluation in a clinical trial.
   * Given that participants undergoing aortic valve replacement are often elderly, multimorbid, and somewhat frail, achieving total and early functional recovery is crucial. Studies in coronary catheterizations have shown better functional recovery and higher quality of life parameters with radial access. No studies have evaluated this in TAVI procedures, and a clinical trial would allow studying this outcome.
   * In conclusion, radial access has emerged as a potentially favorable alternative to femoral access as secondary access in TAVI. Current evidence suggests that radial access may be associated with a lower rate of vascular complications, bleeding, and the need for transfusions, as well as other complications not directly related to access. However, prospective and controlled clinical trials are needed to confirm these findings and establish clear guidelines for choosing secondary access in TAVI. These studies will provide a more accurate and informed understanding of the differences between radial and femoral access in terms of safety and efficacy in the context of TAVI implantation.

EVALUATION OF RELEVANT CLINICAL OUTCOMES:

In addition to vascular complications and other complications, a comparative clinical trial would allow for less biased evaluation of other relevant aspects of the chosen access type, such as radial access feasibility, crossover percentage, procedure success, etc. These results would provide essential information to guide clinical decision-making.

IDENTIFICATION OF BENEFITED PATIENT SUBGROUPS:

A comparative clinical trial could help identify participant subgroups that would benefit more from one type of access over another in terms of clinical outcomes and safety. There are indications of specific predictors of femoral vascular complications, such as peripheral arterial disease, angiographically visualized calcification of the femoral access, chronic kidney disease, etc. These could be verified in such a study, allowing for more personalized care for each participant, optimizing outcomes.

CLINICAL PRACTICE GUIDELINES:

Since evidence in this specific field is scarce and of low quality, the results of a clinical trial would have a significant impact on the development of guidelines and recommendations for clinical practice. Current guidelines provide limited guidance on the choice of secondary access in TAVI. Evidence generated through a clinical trial would help establish more robust and scientifically based recommendations.

In summary, conducting a clinical trial comparing radial and femoral access as secondary access in transfemoral TAVI implantation is essential to fill gaps in existing evidence and provide solid data to support clinical decision-making. This type of trial would allow a systematic assessment of complications, relevant clinical outcomes, and the identification of potentially more benefited participants.

METHODS:

Participants will be randomly assigned to one of two groups: radial access or femoral access. Comprehensive preoperative evaluations will be conducted, including medical history, physical examination, imaging tests, and cardiological assessments. During the TAVI procedure, data on the access used, success, procedure duration, intra-procedural complications, and valve implantation outcomes will be recorded. Results at discharge and 30 days will also be documented.

1. Study Design:

   * A prospective, randomized, controlled clinical trial will be conducted to evaluate radial versus femoral secondary access in percutaneous aortic valve implantation (TAVI). Eligible participants will be randomly assigned to receive radial or femoral access as secondary access in transfemoral TAVI. Data on the access used, success, procedure duration, intra-procedural complications, and valve implantation outcomes will be recorded during the TAVI procedure.
2. Primary Objectives:

   * Compare the overall incidence of major access complications (both vascular and non-vascular) between radial and femoral access at discharge. Major access complications are defined as:
   * Major Vascular Complication:
   * Aortic dissection or rupture.
   * Arterial or venous vascular injury resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or irreversible neurological damage. This includes perforation, dissection, stenosis, ischemia, arterial or venous thrombosis (including pulmonary embolism), arteriovenous fistula, pseudoaneurysm, hematoma, retroperitoneal hematoma, infection, or compartment syndrome.
   * Distal (non-cerebral) embolization from a vascular source resulting in death, amputation, limb or visceral ischemia, or irreversible damage to end organs.
   * Unplanned endovascular or surgical intervention resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or irreversible neurological damage.
   * Device closure failure resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or

   irreversible neurological damage.
   * Major Non-Vascular Complication:
   * Non-vascular or non-cardiac structure perforation, injury, or infection resulting in death, bleeding ≥2 VARC*, irreversible nerve injury, or requiring unplanned intervention or surgical intervention.
   * Device migration, embolization, or malposition resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or irreversible neurological damage.
   * Air or gas embolism resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or irreversible neurological damage.
   * Valve-related infectious endocarditis resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or irreversible neurological damage.
   * Cardiac injury resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or irreversible neurological damage.
   * Valve embolization resulting in death, bleeding ≥2 VARC*, limb or visceral ischemia, or irreversible neurological damage.
3. Secondary Objectives:

   * Compare secondary endpoints between radial and femoral access at discharge and 30 days post-TAVI, including:
   * Individual components of major access complications.
   * Bleeding complications.
   * Transfusions.
   * Peri-procedural renal failure.
   * Stroke.
   * Functional recovery.
   * Quality of life parameters.
4. Study Population:

   * Eligible participants will include adult participants diagnosed with severe aortic stenosis scheduled for elective transfemoral TAVI.
5. Sample Size Calculation:

   * The sample size will be calculated based on the primary endpoint, considering a two-sided significance level of 0.05 and a power of 80%. A presumed major access complication rate of 10% in the femoral group and a hypothesized reduction to 5% in the radial group will be used for the calculation.
6. Statistical Analysis:

   * Descriptive statistics will be used to summarize baseline characteristics. Categorical variables will be compared using chi-square or Fisher's exact test, and continuous variables will be compared using t-tests or non-parametric tests, as appropriate. The primary endpoint will be analyzed using logistic regression, adjusting for relevant covariates. Secondary endpoints will be analyzed similarly. Subgroup analyses will be conducted to explore potential differences in treatment effects across subgroups defined by relevant baseline characteristics.
7. Ethical Considerations:

   * The study will be conducted in accordance with the principles of the Declaration of Helsinki and Good Clinical Practice guidelines. Ethical approval will be obtained from the relevant institutional review board. Informed consent will be obtained from all participants before enrollment.
8. Data Collection and Monitoring:

   * Data will be collected by trained study personnel using standardized case report forms. Data monitoring will be conducted regularly to ensure data quality and participant safety.
9. Trial Oversight:

   * An independent data and safety monitoring board will be established to oversee the progress and safety of the trial. Periodic reviews will be conducted to assess the accumulating data and make recommendations regarding continuation, modification, or termination of the trial.
10. Dissemination of Results:

    * The results of the trial will be disseminated through peer-reviewed publications and presentations at relevant scientific conferences. The data will be shared with the wider scientific community to contribute to the evidence base in the field of TAVI.

EXPECTED OUTCOMES:

This clinical trial aims to provide high-quality evidence regarding the safety and efficacy of radial versus femoral secondary access in transfemoral TAVI. The primary outcome measure, major access complications, will be rigorously assessed, and secondary outcomes will provide a comprehensive understanding of potential differences between the two access types. The results will contribute to the development of evidence-based guidelines and recommendations for clinical practice, ultimately improving participant outcomes and optimizing the delivery of TAVI procedures.

CONCLUSION:

The proposed clinical trial is designed to address the existing gaps in evidence regarding the choice of secondary access in transfemoral TAVI implantation. By conducting a randomized, controlled trial, the investigators aim to provide robust data on the safety and efficacy of radial versus femoral access, informing clinical decision-making and contributing to the development of guidelines in the field of TAVI. This research has the potential to enhance participant care, improve procedural outcomes, and guide future research in the dynamic field of transcatheter aortic valve implantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with severe aortic stenosis and candidates for transfemoral TAVI.
* Secondary access possible through both radial and femoral routes.
* Capacity to provide informed consent.

Exclusion Criteria:

* Specific contraindications for radial or femoral access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-01-08 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
ACCESS RELATED OR BLEEDING COMPLICATIONS | From the enrollment to 4 weeks after the procedure.
  Major and minor access-related complications (VARC-3) and major or greater (VARC ≥2) bleeding complications (BARC)

SECONDARY OUTCOMES:
MACE | From the enrollment to 4 weeks after the procedure.
  Cardiovascular death, stroke or Myocardial infarction requiring revascularization.
bleeding | From the enrollment to 4 weeks after the procedure.
  All bleeding complications and need for red blood transfusions
Quality of life scale | 4 weeks after the procedure
  Quality of life measured by EQ-5D-3L test
Complications not directly TAVI procedure-related | From the enrollment to 4 weeks after the procedure.
  Ex: acute renal failure

IPD SHARING:
Plan to Share IPD: Undecided